CLINICAL TRIAL: NCT05187962
Title: Differential Sensory Block During Labor Epidural Analgesia: a Prospective Observational Study to Investigate the Relationship of Lower and Upper Sensory Block Levels to Cold With Sensory Block to Pinprick and Light Touch
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21-08
Record Dates: First submitted 2021-12-21; First posted 2022-01-12 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Labor Pain
Keywords: sensory block; epidural analgesia; programmed intermittent epidural bolus
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women receiving epidural analgesia for labor: Sensory block level check Patients will have their sensory block level checked using 3 modalities: ice, pin prick and soft touch (cotton ball).

SUMMARY:
Epidural analgesia remains the gold standard for pain control during labor and delivery. Proper assessment of an epidural's level of blockade is important for providing safe and effective analgesia. Previous studies have established that the most commonly tested modality for adequacy of epidural blockade is a patient's sensory blockade to cold temperature. In a study performed at our institution, Soares et. al. (publication pending) documented two thresholds of sensory block to ice: one defined as the lower sensory block level, in which the patient is able to notice the cold sensation but perceives that it is not as cold as a control dermatome; the other defined as the upper sensory block level, in which the patient perceives that the cold sensation is at approximately the same temperature as if it were applied to a non-anesthetized area such as the neck or face. Although this a known finding to nurses and physicians assessing the sensory block to ice, this phenomenon and its magnitude has not been previously reported in epidural anesthesia. The goal of this study is to examine patients with labour epidurals and to determine the dermatomal relationship between the lower and upper sensory block levels to cold when compared with sensory blockade to both pinprick and light touch.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status Classification II and III parturients
* Requested and received a labour epidural
* Capable of consenting to the study
* Have no language barrier which may obfuscate the sensory block assessment
* Are receiving programmed intermittent epidural boluses (PIEB) for maintenance analgesia, which is the Mount Sinai Hospital default maintenance regimen

Exclusion Criteria:

* Medical comorbidities that could compromise the body's sensitivity to cold, pinprick, or touch
* Epidurals performed under a combined spinal-epidural (CSE) or dural puncture epidural (DPE) technique
* Epidurals with a documented unintentional dural puncture
* Inadequate epidural analgesia requiring either manually administered epidural boluses, an increase in the concentration of their maintenance local anesthetic, or a repeat of their epidural

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Women admitted to the Labor and Delivery unit at Mount Sinai Hospital that receive epidural analgesia for labour.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Lower sensory block level: ice test | 5 minutes
  The lower sensory block level to ice, defined as the dermatome at which there is a complete loss of cold perception.
Upper sensory block level: ice test | 5 minutes
  The upper sensory block level to ice is defined as the dermatome at which there is an altered cold perception without complete sensitivity loss.
Lower sensory block level: pinprick test | 5 minutes
  The lower sensory block level to pinprick, defined as the dermatome at which there is a complete loss of sharp sensation.
Upper sensory block level: pinprick test | 5 minutes
  The upper sensory block level to pinprick is defined as the dermatome at which there is an altered sharp sensation without complete sensitivity loss.
Sensory block level: soft touch test | 5 minutes
  The sensory block level using soft touch is defined as the dermatome below which the patient can feel a light touch.

SECONDARY OUTCOMES:
Motor block score using Bromage score | 5 minutes
  Motor block will be assessed with the Bromage score: 0 = able to raise the extended leg; 1 = unable to raise the extended leg but able to flex knees; 2 = unable to flex knees, but able to flex ankle; 3 = unable to flex ankle.

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casellato JF, Balki M, Wang A, Ye XY, Downey K, Carvalho JCA. Differential sensory block during labour epidural analgesia: a prospective observational study to investigate the relationship of lower and upper sensory block levels to cold, pinprick, and light touch. Can J Anaesth. 2024 Jun;71(6):802-807. doi: 10.1007/s12630-023-02638-5. Epub 2024 Jan 30. PMID 38291174